CLINICAL TRIAL: NCT03676153
Title: Assessing the Impact of an Integrative Care Training Program for Nurses in Manual Therapies, Relaxation, Lifestyle Changes and Traditional Medicine on Quality of Life in Oncology Patients: A Randomized Controlled Study
Brief Title: Integrative Care Training Program for Nurses on Supportive Cancer Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Eran Ben-Arye, Medical Director, Integrative Oncology Program, Oncology Service, Lin and Carmel Medical Centers, Carmel Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMC-18-0139-CTIL
Record Dates: First submitted 2018-09-13; First posted 2018-09-18 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Cancer; Quality of Life; Nurse's Role
Keywords: Integrative medicine; Supportive and Palliative care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Pragmatic study examining the impact of a nurse-guided self-administered integrative medicine intervention on quality-of-life outcomes in cancer care.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nurse-guided arm (Experimental): Nurse-provided guidance following an integrative medicine treatment program, for patient implementation of self-administered manual therapies, relaxation, lifestyle changes and traditional medicine.
  Interventions: Other: Nurse-provided guidance; Other: Integrative medicine treatment program
- Non nurse-guided arm (Active Comparator): Integrative medicine treatment program, with no nurse-provided guidance on patient implementation of self-administered manual therapies, relaxation, lifestyle changes and traditional medicine.
  Interventions: Other: Integrative medicine treatment program

INTERVENTIONS:
Other: Nurse-provided guidance — Nurse-provided guidance following an integrative medicine treatment program, for patient implementation of self-administered manual therapies, relaxation, lifestyle changes and traditional medicine.
  Arms: Nurse-guided arm
Other: Integrative medicine treatment program — Integrative medicine treatment program

SUMMARY:
The integration of complementary medicine in supportive and palliative cancer care (i.e., Integrative Oncology) is becoming more prevalent in many of the leading oncology centers in Israel and worldwide. Guidelines for these practices, as established by the Society for Integrative Oncology, were adopted in 2018 by the American Society of Clinical Oncology.

The proposed study will be conducted within a pragmatic, randomized and controlled format, and will examine the impact of a nurse-guided intervention on 540 oncology patients undergoing Integrative Oncology treatments for quality of life (QOL)-related concerns during adjuvant/neo-adjuvant or curative/palliative treatments. Patients in both study arms will undergo patient-tailored integrative treatments, which will include manual and relaxation therapies, acupuncture and lifestyle changes. The integrative treatments will be provided by trained integrative oncology practitioners. Patients in the intervention arm of the study will receive additional nurse-guided instruction in the self-administration of manual therapies, relaxation, lifestyle changes and traditional medicine practices.

DETAILED DESCRIPTION:
The integration of complementary medicine in supportive and palliative cancer care (i.e., Integrative Oncology) is becoming more prevalent in many of the leading oncology centers in Israel and worldwide. Guidelines for these practices, as established by the Society for Integrative Oncology, were adopted in 2018 by the American Society of Clinical Oncology.

The proposed study will be conducted within a pragmatic, randomized and controlled format, and will examine the impact of a nurse-guided intervention on 540 oncology patients undergoing Integrative Oncology treatments for quality of life (QOL)-related concerns during adjuvant/neo-adjuvant or curative/palliative treatments. Patients in both study arms will undergo patient-tailored integrative treatments, which will include manual and relaxation therapies, acupuncture and lifestyle changes. The integrative treatments will be provided by trained integrative oncology practitioners. Patients in the intervention arm of the study will receive additional nurse-guided instruction in the self-administration of manual therapies, relaxation, lifestyle changes and traditional medicine practices.

The primary study outcome will be the assessment of the impact of the integrative treatment (with vs. without the nurse-guided intervention) on patient QOL-related concerns, from baseline to 48 hours following the intervention. For this purpose, two patient-reported outcome measures (PROMs) will be administered: the Edmonton Symptom Assessment Scale (ESAS) and the Measure Yourself Concern and Wellbeing (MYCAW) questionnaire. Secondary outcome measures will include the need for medications for supportive/palliative care-related indications (pain, nausea, anxiety/depression, constipation/diarrhea, etc.); and the rates of referral of patients to the services provided by the supportive/palliative care service.

ELIGIBILITY:
Inclusion Criteria:

* Oncology patients undergoing treatment within an adjuvant, neo-adjuvant, curative or palliative setting.

Exclusion Criteria:

* Patients who are unable to sign informed consent
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-03-20 (Actual)

PRIMARY OUTCOMES:
Measure Yourself Concerns and Wellbeing (MYCAW) | 48 hours
  Scale from 0 (not bothering me at all) to 6 (bothers me greatly)

SECONDARY OUTCOMES:
Edmonton Symptom Assessment Scale (ESAS) | 24 hours
  Scale from 0 (no symptom) to 10 (worst possible symptom)

CONTACTS AND LOCATIONS:
Locations (1):
- Lin Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ben-Arye E, Shulman B, Eilon Y, Woitiz R, Cherniak V, Shalom Sharabi I, Sher O, Reches H, Katz Y, Arad M, Schiff E, Samuels N, Caspi O, Lev-Ari S, Frenkel M, Agbarya A, Admi H. Attitudes Among Nurses Toward the Integration of Complementary Medicine Into Supportive Cancer Care. Oncol Nurs Forum. 2017 Jul 1;44(4):428-434. doi: 10.1188/17.ONF.428-434. PMID 28632238
- [Derived] Ben-Arye E, Tapiro Y, Baruch R, Tal A, Shulman B, Gressel O, Israeli P, Dagash J, Yosipovich A, Shalom Sharabi I, Zimmermann P, Samuels N. Integrative oncology for palliative care nurses: pre-post training evaluation. BMJ Support Palliat Care. 2024 May 17;14(2):178-182. doi: 10.1136/spcare-2022-004117. PMID 36690415